CLINICAL TRIAL: NCT05930756
Title: A Randomized Controlled Trial Comparing the Efficacy of a Three-Point Versus a Six-Point Genicular Nerve Radiofrequency Ablation for Chronic Knee Osteoarthritis
Brief Title: 3-point vs 6-point GNRFA for Chronic KOA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GNRFA 2023
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis, Knee; Chronic Pain
Keywords: Radiofrequency ablation; Osteoarthritis, Knee; Genicular radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient will be sedated and positioned so that they will not know which of the two treatments they receive. The outcomes assessor will not know which treatment the patient received, as they will not be present during the procedure. The care provider (if present) will not be told. Only care providers involved in the procedure are unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-target GNRFA technique (T1) (Active Comparator): Radiofrequency ablation will target three of the genicular nerves: the superolateral genicular nerve, the superomedial genicular nerve, and the inferomedial genicular nerve.
  Interventions: Procedure: Radiofrequency ablation
- Six-target GNRFA technique (T2) (Active Comparator): Radiofrequency ablation will target six of the genicular nerves: the superolateral genicular nerve, the superomedial genicular nerve, the inferomedial genicular nerve, two branches from the nerve of vastus intermedius, and the recurrent fibular nerve
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Genicular radiofrequency ablation uses thermal energy to percutaneously create lesions in neural tissues of the genicular nerves that innervate the anterior knee capsule and disrupt the conduction of pain signals.

SUMMARY:
The goal of this clinical trial is to compare three-point and six-point Genicular Nerve Radiofrequency Ablation (GNRFA) in adults with chronic knee osteoarthritis (KOA). The main question it aims to answer is whether six- target GNRFA technique is more efficacious than standard three-target GNRFA technique in managing the pain and function of KOA. Consented patients who respond to a diagnostic block will be randomly assigned to either three-point or six-point GNRFA. Researchers will compare pain and function in these two groups.

DETAILED DESCRIPTION:
Background Knee osteoarthritis (KOA) is a leading cause of chronic knee pain and disability, with a lifetime prevalence of 45%1. While treatment for symptomatic KOA includes physical therapy, oral anti-inflammatory medications and intra-articular steroid injections, the definitive treatment is total knee arthroplasty. However, approximately 600 000 fewer surgeries were performed in the first three months of the COVID pandemic which has created an overwhelming backlog of patients awaiting elective surgical management2. The significant delays caused by the backlog in surgery are leading to worsened pain requiring increased opioid use, functional impairment, and psychological well-being of patients3. Therefore, the use of fluoroscopy-guided genicular nerves radiofrequency ablation (GNRFA) has become a valuable treatment option for patients either awaiting arthroplasty or are ineligible for arthroplasty due to comorbidities or for personal preference3.

GNRFA uses thermal energy to percutaneously create lesions in neural tissues of the genicular nerves that innervate the anterior knee capsule and disrupt the conduction of pain signals. Classically, the three branches of the genicular nerve that are targeted in this procedure include the superolateral genicular nerve (SLGN), superomedial genicular nerve (SMGN) and the inferomedial genicular nerve (IMGN). As these nerves run consistently on their way to the joint between the diaphysis and metaphysis of the femur and tibia, they provide reliable landmarks to targets for an RFA procedure7. Subsequently, the safety of GNRFA in the management of KOA and its greater efficacy compared to other options including intraarticular steroid injections, viscosupplementation and oral analgesics has been replicated in several large clinical studies and systematic reviews, leading to its wide adoption1,4-7. The knee joint innervation is much more extensive, however, as 10 nerves innervate the knee capsule. Unfortunately, not all of them can be targeted percutaneously8. Recent anatomic validation studies, though, have revealed three additional nerves that are suitable targets under fluoroscopy with bony landmarks. These include the two branches from the nerve of vastus intermedius (VIN), which run consistently in the lateral and medial third of the femoral diaphysis 2 cm above the patella, and the recurrent fibular nerve (RFN), which runs consistently on the surface of the fibular head at its widest diameter. Consequently, a six-target technique has been described that includes the recurrent fibular nerve (RFN), and the two branches of the VIN in addition to the conventional three targets9,10.

To date, four-, and six-target knee neurolysis procedures have shown to be effective pain relief in KOA, showing significant improvement in validated pain and functional scores for more than 6 months after the procedure11-14. However, the studies demonstrating these results have primarily consisted of case series with small sample sizes11,13. Thus far, only a four-target technique (adding a single lesion above the patella) has been retrospectively investigated against the original three-target technique, showing improvement in pain in both groups with less opiate medications consumption in the four target group12. Therefore, targeting additional nerves to the three-target technique may improve pain and functional outcomes for this relatively new procedure which has become particularly valuable in the last decade to manage pain due to knee OA and especially during the covid 19 pandemic, where the waiting list of patients for joint replacement has been significantly increasing.

Purpose The overall purpose of this randomized controlled trial is to evaluate the efficacy of a six- target GNRFA technique (T2) in managing the pain and function of KOA patients in comparison to the standard three-target GNRFA technique (T1).

Specific Aims:

To compare the change in Western Ontario and McMaster Universities Arthritis (WOMAC) scores from baseline at 12 weeks compared between T1 and T2 To compare the change in patient-reported pain scale (NRS) between T1 and T2 To compare change in oral opioid intake in morphine equivalents between T1 and T2 To compare the percentage of patients who have improved pain and function between T1 and T2 To assess the population characteristics of patients that have improved outcomes when treated with T1 and T2 including laterality, body mass index, age, comorbidities, degree of KOA, medications, smoking status, and any adverse effects.

To assess the safety and side effect profile of T1 and T2

Patients identified from the clinic booking list referred for suitability of GNRFA from orthopedic surgeons will be approached at the EEPC. Once deemed eligible, after discussion of the therapeutic options and potential benefits and risk of GNRFA by a pain physician, a research assistant (RA) will approach patients for study inclusion and obtain informed consent. Patients who have offered consent will be assessed for baseline scores of WOMAC, NRS and analgesic intake. They will then undergo a diagnostic block in which they receive a Lidocaine (0.5 mL of 2%) injection at the SLGN, SMGN and IMGN under ultrasound guidance. If patients report an improvement in NRS pain score by 50% at 20 minutes, they will be included as a subject to be randomly assigned to one of the GNRFA treatment schedules, three- (T1) or six-target (T2).

Sample Size, Recruitment Rate The following sample size estimates were calculated based on a two-sided alpha=5%, and power=80%. Based on the study by Sari et. al16, the mean change in WOMAC scores from baseline were varied between 5-10 and SDs for both groups were varied between 9-12. Calculations were determined using WinPepi Software (Version 11.65). Sample size estimates adjusted for non-inclusion (ineligibility) has also been presented.

Based on this sample size estimation, we have determined the sample size to be 80 (40 in each arm), adjusting for 30% non-inclusion.

The recruitment rate is expected to take 8-12 months at a rate of approximately 3-5 patients per week which is a feasible rate determined by our currently ongoing retrospective study comparing T1 and T2.

Randomization/Allocation and Blinding Patients who responded to the diagnostic block will subsequently be given unique number identifiers and assigned to each arm in a 1:1 allocation ratio using computer-generated block randomization. These patients will be identified in the anesthesia chart. The pain physician performing the interventional procedures will be provided the assigned treatment arm of each subject in an encrypted USB key prior to performing the subjects' assigned treatments. Patients, data collectors and analysts will be blinded. Pain physician will not be blinded given the nature of this study.

Study Interventions After confirming the unique number identifier, the radiofrequency will be performed on the day of surgery, in a designated operating room at St Joseph's Hospital, king campus. Intravenous (IV) access will be established, and standard monitoring will be applied including non-invasive blood pressure, electrocardiogram, and pulse oximetry. Sedation and anxiolytics may be used as clinically appropriate by the pain doctor performing the procedure. The radiofrequency will be performed by one of the three pain doctors from the study group as they have received extensive training and experience performing the procedure. The patient will be placed in a supine position, and the index knee is flexed 30 degrees using a bolster, which will facilitate a clear lateral view of the knee. The area over the knee will be sterilized with disposable swabs of 2% chlorhexidine in 70% isopropyl alcohol and then draped in a sterile fashion. After prepping and draping the knee, fluoroscopic scout images will be used to align the tibial plateau in a true anterior-posterior (AP) view.

T1: A skin wheal will be placed at the superomedial and superolateral of the knee where the diaphysis joins metaphysis of the femur and in the inferomedial side of the knee where the diaphysis and metaphysis tibia join. Three mL of 1% lidocaine will be administered to anesthetize the skin and neighboring subcutaneous tissues. Then, a 22 G spinal needle will be used to enter the skin wheal and walk off from periosteum, depositing an additional 3 mL of lidocaine 1% on each of the three sites to anesthetize deep tissues before the radiofrequency needle insertion. Then an 18 G 1 cm uninsulated curve radiofrequency needle will be advanced through the skin wheal at each of the three sites until it contacts the periosteum of the superomedial, superolateral knee femur and the inferomedial knee tibia. A true lateral fluoroscopic view will then be obtained by superimposing the femoral condyles. Each needle will be advanced until they reach the posterior third of the femur at the superomedial and superolateral knee sites and the posterior third of the tibia at the inferomedial knee site. Then continuous radiofrequency for 90 seconds at 80 degrees will be applied. The three needles will then be moved anteriorly until they reach the middle third of the femur and tibia respectively. Another continuous radiofrequency lesion will be applied with same parameters. Finally, the three needles will be moved anteriorly until they reach the anterior third of the femur and tibia respectively. An additional lesion will be created using same parameters. Then before removing the needles, 3 mL of Bupivacaine 0.5% will be administered for postoperative pain control through each needle.

T2: In addition to receiving the T1 intervention, the T2 arm will also receive lesions to the lateral and medial branches of the nerve of vastus intermedius. A True AP view will be obtained as previously described. A skin wheal will be placed 2 cm above the upper pole of patella at the medial third (medial branch of vastus intermedius) and lateral third (lateral branch of vastus intermedius) of the femur. One mL of lidocaine 1% will be injected on each site to anesthetize skin and surrounding subcutaneous tissues. Then an 18 g 1 cm uninsulated curve radiofrequency needle will be advanced through each skin wheal until reaching periosteum. Then continuous radiofrequency will be applied using 80 degrees for 90 seconds. The radiofrequency needles will be repositioned 5 mms apart from the first lesion, and another continuous radiofrequency will be applied using same parameters to ensure lesioning the whole area of the medial and lateral third of the femur, where the nerve runs from caudally. Before removing the needles, 1 mL of bupivacaine 0.5% will be administered through each needle.

Finally, the recurrent fibular nerve will be targeted. True AP views will be obtained as previously described. A skin wheal will be placed 0.5-1 cm lateral ti the lateral tibial condyle at the cranio-caudal level of the lower third of the fibular head. One mL of 1% lidocaine will be administered to anesthetize the skin and neighboring subcutaneous tissues. The radiofrequency needle will then be advanced through the skin wheal. From this slightly lateral entry point, the needle will be advanced until it meets the periosteum of the lateral tibial condyle. Then the needle tip is positioned at the cranio-caudal level of the lower third of the fibular head (widest aspect of fibular head) avoiding periosteum contact until final advancement. A true lateral fluoroscopic view will then be obtained as described before, and the needle tip will be repositioned 1-2 mm anterior to the fibular head. Distance from radiofrequency lesion to skin may be enhanced by lifting the skin away from the periosteum using additional local anesthetic (following motor testing). Motor testing is performed at 2HZ and 2 mV to ensure enough distance from the fibular nerve. Then 1 mL of lidocaine 1% will be administered to anesthetize the recurrent fibular nerve. The continuous radiofrequency will be applied using 80 degrees for 60 seconds. Then the needle will be slightly removed and 1 mL of bupivacaine 0.5% administered for post operative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Chronic knee pain for at least 3 months with radiological evidence of KOA graded 2-4 on the Kellgren-Lawrence scale as determined by a radiologist

Exclusion Criteria:

* unwilling,
* unable to communicate in English,
* have acute knee pain,
* prior knee surgery,
* allergies to local anesthetics,
* chronic opioid consumption of daily morphine equivalent of >30 mg for at least four weeks prior to procedure,
* neurologic diseases affecting the lower limbs (i.e. previous CVA, MS),
* connective tissue diseases affecting the knee,
* treatment with intra-articular steroid injections and/or hyaluronic acid in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale score | 12 weeks
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale quantifies knee pain severity with activities of daily living. It is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Higher points signify higher levels of functional difficulty. This will be captured by change in WOMAC scores from baseline at 12 weeks

SECONDARY OUTCOMES:
Numerical rating scale | 4 time points: 30 min, 4 weeks, 12 weeks, 24 week spost procedure
  Patient-reported 11-point scale where 0 is no pain and 10 the worst pain imaginable, at rest and walking
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale score | 2 time points: 4 weeks and 24 weeks post procedure
  The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale quantifies knee pain severity with activities of daily living. It is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items). Higher points signify higher levels of functional difficulty.
Opioid intake | 24 weeks post procedure
  Calculated as total morphine equivalents

OTHER OUTCOMES:
Incidence of adverse effects | 3 time points: 4 weeks, 12 weeks, and 24 weeks post procedure
  Patients will be asked about adverse events such as motor dysfunction, burning pain in dermatomal distribution, localized burning pain, infection, and haematoma

REFERENCES:
- [Background] Conger A, Gililland J, Anderson L, Pelt CE, Peters C, McCormick ZL. Genicular Nerve Radiofrequency Ablation for the Treatment of Painful Knee Osteoarthritis: Current Evidence and Future Directions. Pain Med. 2021 Jul 25;22(Suppl 1):S20-S23. doi: 10.1093/pm/pnab129. PMID 34308957
- [Background] Molloy, L. (2022, May 10). Wait times for priority procedures in Canada. CIHI. Retrieved September 10, 2022, from https://www.cihi.ca/en/wait-times-for-priority-procedures-in-canada
- [Background] Oudhoff JP, Timmermans DR, Knol DL, Bijnen AB, van der Wal G. Waiting for elective general surgery: impact on health related quality of life and psychosocial consequences. BMC Public Health. 2007 Jul 19;7:164. doi: 10.1186/1471-2458-7-164. PMID 17640382
- [Background] Tate, Q., Conger, A., Burnham, T. et al. The Effectiveness and Safety of Genicular Nerve Radiofrequency Ablation for the Treatment of Recalcitrant Knee Pain Due to Osteoarthritis: a Comprehensive Literature Review. Curr Phys Med Rehabil Rep 7, 404-413 (2019). https://doi.org/10.1007/s40141-019-00246-3
- [Background] Fogarty AE, Burnham T, Kuo K, Tate Q, Sperry BP, Cheney C, Walega DR, Kohan L, Cohen SP, Cushman DM, McCormick ZL, Conger A. The Effectiveness of Fluoroscopically Guided Genicular Nerve Radiofrequency Ablation for the Treatment of Chronic Knee Pain Due to Osteoarthritis: A Systematic Review. Am J Phys Med Rehabil. 2022 May 1;101(5):482-492. doi: 10.1097/PHM.0000000000001813. Epub 2021 May 27. PMID 35006653
- [Background] Hong T, Wang H, Li G, Yao P, Ding Y. Systematic Review and Meta-Analysis of 12 Randomized Controlled Trials Evaluating the Efficacy of Invasive Radiofrequency Treatment for Knee Pain and Function. Biomed Res Int. 2019 Jun 26;2019:9037510. doi: 10.1155/2019/9037510. eCollection 2019. PMID 31346525
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] McCormick ZL, Cohen SP, Walega DR, Kohan L. Technical considerations for genicular nerve radiofrequency ablation: optimizing outcomes. Reg Anesth Pain Med. 2021 Jun;46(6):518-523. doi: 10.1136/rapm-2020-102117. Epub 2021 Jan 22. PMID 33483425
- [Background] Tran J, Peng PWH, Lam K, Baig E, Agur AMR, Gofeld M. Anatomical Study of the Innervation of Anterior Knee Joint Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 May;43(4):407-414. doi: 10.1097/AAP.0000000000000778. PMID 29557887
- [Background] Fonkoue L, Stoenoiu MS, Behets CW, Steyaert A, Kouassi JK, Detrembleur C, Cornu O. Validation of a new protocol for ultrasound-guided genicular nerve radiofrequency ablation with accurate anatomical targets: cadaveric study. Reg Anesth Pain Med. 2021 Mar;46(3):210-216. doi: 10.1136/rapm-2020-101936. Epub 2020 Dec 3. PMID 33273065
- [Background] Ahmed A, Arora D. Ultrasound-Guided Neurolysis of Six Genicular Nerves for Intractable Pain from Knee Osteoarthritis: A Case Series. Pain Pract. 2019 Jan;19(1):16-26. doi: 10.1111/papr.12710. Epub 2018 Aug 8. PMID 29761638
- [Background] Koshi E, Meiling JB, Conger AM, McCormick ZL, Burnham TR. Long-term clinical outcomes of genicular nerve radiofrequency ablation for chronic knee pain using a three-tined electrode for expanded nerve capture. Interv Pain Med. 2021 Nov 19;1(1):100003. doi: 10.1016/j.inpm.2021.100003. eCollection 2022 Mar. PMID 39301447